CLINICAL TRIAL: NCT01919320
Title: SynCardia Companion 2 Driver System Post Approval Study Protocol With INTERMACS™-Based Data Collection
Acronym: C2 PAS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: SynCardia Systems. LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: RA-409; Data Collection via INTERMACS (Registry Identifier: INTERMACS Registry)
Record Dates: First submitted 2013-08-06; First posted 2013-08-09 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Bi-ventricular Failure
Keywords: SynCardia; Total Artificial Heart; TAH-t

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- CSS Console TAH-t Patients: All TAH-t patients implanted while supported with the CSS Console who were enrolled in the INTERMACS Registry and implanted with the TAH-t on or after June 20, 2012.
  Interventions: Device: CSS Console TAH-t Patients
- C2 Driver System TAH-t Patients: 200 TAH-t patients implanted while supported by the Companion 2 (C2) Driver System who were enrolled in the INTERMACS Registry and implanted with the TAH-t on or after June 20, 2012.
  Interventions: Device: C2 Driver System TAH-t Patients
- All TAH-t Patient Records: All records for TAH-t patients enrolled in the INTERMACS Registry will be reviewed to support Objective 2 of the protocol.
  Interventions: Device: C2 Driver System TAH-t Patients; Device: CSS Console TAH-t Patients

INTERVENTIONS:
Device: C2 Driver System TAH-t Patients — Comparison of two pneumatic drivers supporting the SynCardia TAH-t
  Other Names: SynCardia
  Groups: All TAH-t Patient Records; C2 Driver System TAH-t Patients
Device: CSS Console TAH-t Patients — Comparison of two pneumatic drivers supporting the SynCardia TAH-t.
  Other Names: SynCardia
  Groups: All TAH-t Patient Records; CSS Console TAH-t Patients

SUMMARY:
Study Purpose

The purpose of this PAS is to confirm that patients implanted with the temporary Total Artificial Heart (TAH-t) and supported with the Companion 2 Driver System have outcomes similar to those patients implanted with the TAH-t and supported with the CSS Console. The data collection mechanism for this study is the INTERMACS Registry.

Study Objectives

Primary Objective 1:

To confirm that patients implanted with the TAH-t and supported by the Companion 2 Driver System have outcomes similar to those patients implanted with the TAH-t and supported by the CSS Console.

Primary Objective 2:

To compare positive outcome rates for all TAH-t patients entered in the Intermacs Registry initially supported with the Companion 2 Driver System to positive outcome rates for all TAH-t patients initially supported by the CSS Console.

Primary Objective 3:

To review additional data (patient survival, adverse event rates and bridge to transplant rates) to support the conclusion that the use of an artificial heart is reasonable and necessary for the treatment of irreversible biventricular failure in Medicare/Medicaid patients.

Secondary Objective:

* To evaluate the incidence of adverse events (AEs). The AEs will follow the definitions in the INTERMACS Registry.

Study Hypothesis: Primary Objective 1 The primary hypothesis is that the positive outcome rate (defined as transplant , transfer to the Freedom Driver System support, or continuing on implant driver support, whichever occurs first; assessed at three and six months post-implant) for patients supported with the Companion 2 Driver System is non-inferior to the survival rate for patients supported with the Circulatory Support System (CSS) Console.

Data Collection The data will be collected as defined in the INTERMACS Protocol and the patients will be followed at one week, one month, three months and six months or until their study endpoint is reached.

Data Analysis

Primary Objective 1:

Data analysis will provide descriptive statistics on enrollment, adverse events, and outcomes for TAH-t patients who were implanted while supported with the Companion 2 Driver System compared to TAH-t patients who were implanted while supported with the CSS Console.

Primary Objective 2:

Data analysis will provide descriptive statistics on enrollment, adverse events, and outcomes for all TAH-t patients enrolled in the INTERMACS Registry.

Phase I as described above was completed; Phase II of Study design is under review by FDA with anticipated initiation in early 2021.

ELIGIBILITY:
Inclusion Criteria:

* Implanted with the TAH-t
* Patient or their legal representative has signed an informed consent (ICF) form for INTERMACS Registry participation or waiver of consent has been approved at the implanting institution.

Exclusion Criteria:

* Patient or legal guardian has not signed an ICF for INTERMACS Registry participation, if required at the institution.
* Patient is incarcerated.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with bi-ventricular failure at risk of imminent death who are implanted with the SynCardia temporary Total Artificial Heart (TAH-t) AND who have enrolled in the INTERMACS Registry
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-12; Primary Completion 2022-12 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Positive outcome rates at three months and six months Post TAH-t Implant (Concurrent Cohort) | Three and Six Months Post-TAH-t Implant
  The positive outcome rates, defined as transplant, transfer to the Freedom Driver System, or continuing on implant driver support (whichever occurs first) for patients implanted on or after June 20, 2012 and supported with the Companion 2 Driver System will be compared to the positive outcome rates at three and six months for patients implanted on or after June 20, 2012 and supported with the Circulatory Support System (CSS) Console.
  The analysis will include a lower one-sided 95% confidence bound on the observed survival rate for patients supported with the Companion 2 Driver system which will be compared to the CSS Console survival rate to evaluate non-inferiority.
Positive outcome rates at three months and six months Post TAH-t Implant (Cumulative Cohort) | Three and Six Months Post-TAH-t Implant
  The positive outcome rates, defined as transplant, transfer to the Freedom Driver System, or continuing on implant driver support (whichever occurs first) for patients supported with the Companion 2 Driver System will be compared to the positive outcome rates at three and six months for patients supported with the Circulatory Support System (CSS) Console.
  The analysis will include a lower one-sided 95% confidence bound on the observed survival rate for patients supported with the Companion 2 Driver system which will be compared to the CSS Console survival rate to evaluate non-inferiority.

SECONDARY OUTCOMES:
Review of all TAH-t patient records in the INTERMACS Registry to confirm acceptability of treatment for bi-ventricular failure. | Three and Six Months Post-TAH-t Implant
  To review additional data (patient survival, adverse event rates and bridge to transplant rates) to support the conclusion that the use of an artificial heart is reasonable and necessary for the treatment of irreversible biventricular failure as ordered by the CMS National Coverage Decisions which requires enrollment of Medicare patients in approved studies for evidence development.

OTHER OUTCOMES:
Comparison of Adverse Event Rates | Three and Six Months Post-TAH-t Implant or Study Endpoint, whichever occurs first.
  To evaluate the incidence of adverse events (AEs). The AEs will follow the definitions in the INTERMACS Registry.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Arabia, MD, Principal Investigator — Banner University Medical Center